CLINICAL TRIAL: NCT04705597
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Investigate the Efficacy and Safety of BGE-175 in Hospitalized Adults With COVID-19
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of BGE-175 in Hospitalized Adults With Coronavirus Disease 2019 (COVID-19) That Are Not in Respiratory Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The incidence of COVID-19 hospitalization cases decreased to a level that continued enrollment was no longer feasible
Sponsor: BioAge Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGE-175-201
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: COVID-19; BGE-175; BioAge; Respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — asapiprant

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGE-175 (Experimental): BGE-175 tablet to be taken by mouth once a day for 14 days
  Interventions: Drug: BGE-175
- Placebo (Placebo Comparator): Placebo tablet to be taken by mouth once a day for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BGE-175 — Drug
  Arms: BGE-175
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and efficacy of BGE-175 in participants ≥ 50 years of age hospitalized with documented COVID-19.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel-group, multicenter, double-blind study of BGE-175 administered PO or NG in participants ≥ 50 years of age and hospitalized with documented COVID-19 who are not yet in respiratory failure.

After signing informed consent, participants will be screened upon presentation at the hospital. Screening will include full physical examination, vital signs, safety laboratory evaluation, oxygen saturation, pre-diagnostics to measure prostaglandin D2 (PGD2) status, and baseline assessment of World Health Organization (WHO) Ordinal Scale for COVID-19. If confirmed that the participant qualifies for this protocol according to listed inclusion and exclusion criteria, participants will receive the first dose of study medication, PO. The participant will then receive study medication PO or NG (if intubated or unable to swallow medication) once daily, at approximately the same time each day for up to 13 additional days. Study medication will be administered in addition to standard of care deemed appropriate by the treating physician(s). Participants will be randomized to receive BGE-175 or placebo. Participants will be monitored daily for all relevant efficacy outcomes, oxygen saturation, and adverse events. Blood will be drawn periodically for safety laboratory measurements, plasma kinetics, lymphocyte subsets, C-reactive protein, and cytokines. Nasopharyngeal swabs will be collected to measure viral load. Participants will be monitored for 14 days after administration of the last dose (Day 28) and followed through Day 57.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide informed consent that is documented per local requirements
* An understanding, ability, and willingness to fully comply with study procedures and restrictions
* Hospitalized subjects with a confirmed SARS-CoV-2 infection
* Laboratory (polymerase chain reaction [PCR]) confirmed infection with SARS-CoV-2
* Age ≥ 50 years
* COVID-19 illness of any duration, and oxygen saturation measurements ≤ 94% over 5 minutes on room air (Note: low flow oxygen is permitted, but room air oxygen saturation must be ≤ 94%)
* Not in respiratory failure as defined by at least one of the following:

  1. Respiratory failure defined by requiring at least one of the following:

     * Endotracheal intubation and mechanical ventilation
     * Oxygen delivered by high-flow nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5)
     * NIPPV
     * ECMO
     * Clinical diagnosis of respiratory failure (i.e., need for one of the preceding therapies, but preceding therapies are not being administered because it is unavailable in the current setting)
  2. Hemodynamic compromise (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg) or requiring vasopressors
  3. Multi-organ dysfunction/failure
* Females subjects of childbearing potential must have a negative pregnancy test at screening or pre-treatment on Day 1
* Male and female subjects of childbearing potential must agree to use methods of contraception that are consistent with local regulations for those participating in clinical studies

Exclusion Criteria:

* Participation in any other randomized, controlled clinical trial of an experimental treatment for COVID-19 (uncontrolled, compassionate use trials are allowed)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Currently participating in a vaccination trial for SARS-CoV-2
* Known positive test for influenza A or influenza B at the time of screening
* Positive for human immunodeficiency virus (HIV) that is not controlled with current treatment
* Hepatitis B surface antigen, or Hepatitis C positive at the time of screening. Subjects who are positive for Hepatitis C but have Hepatitis C virus (HCV) RNA below the limit of quantitation may be enrolled. Subjects with Hepatitis B, but with undetectable viral load, may be enrolled.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × the upper limit of normal (ULN)
* Stage 4 severe chronic kidney disease (i.e., estimated glomerular filtration rate [eGFR] < 30 mL/min) or acute renal failure resulting in eGFR < 30 mL/min
* Serious comorbidity, including:

  1. Myocardial infarction (within the last month)
  2. Moderate or severe heart failure (New York Heart Association [NYHA] class III or IV)
  3. Acute stroke (within the last month)
  4. Uncontrolled malignancy. Uncontrolled malignancy would include cancers that are not considered in remission, or solid tumor or hematological malignancies with evidence of disease progression in the past 3 months (i.e., there is evidence of disease progression by Response Evaluation Criteria in Solid Tumours [RECIST] or equivalent relevant criterion for the type of malignancy), and are not considered effectively managed with ongoing treatment as determined by the investigator
  5. Recent severe thromboembolic disease or evidence of severe thromboembolic disease defined as a current large vessel thromboembolic event or a thromboembolic event within the past 3 months (e.g., deep vein thrombosis [DVT], pulmonary embolism, ischemic stroke, transient ischemic attack) requiring interventional treatment. This exclusion does not prohibit prophylaxis for thromboembolic events, including those considered possible with concurrent SARS-CoV-2 infection.
* History of severe allergic or anaphylactic reactions or hypersensitivity to the study drug
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive study treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Wilkerson, MD, Principal Investigator — University of Maryland, Baltimore
Locations (26):
- United States (11):
  - Banner Health, Mesa, Arizona
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Long Beach Medical Center, Long Beach, California
  - UCI Center for Clinical Research, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - North Colorado Medical Center, Greeley, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - University of Florida - Health, Jacksonville, Jacksonville, Florida
  - Baptist Health, Lexington, Lexington, Kentucky
  - University of Maryland Medical System, Baltimore, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
- Argentina (3):
  - Clinica Privada Independencia, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Sanatorio De La Trinidad Mitre, Buenos Aires, Buenos Aires F.D.
  - Clinica Adventista Belgrano (CAB), Buenos Aires, Buenos Aires F.D.
- Brazil (12):
  - Hospital Universitário Cassiano Antônio de Moraes, Vitória, Espiritu Santo
  - Hospital Felicio Rocho (HFR), Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Hospital Ana Nery Santa Cruz do Sul, Santa Cruz do Sul, Rio Grande Do Sol
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Clínica Supera Oncologia, Chapecó, Santa Catarina
  - Unidade de Pesquisa Clinica da Fundação Pio XII - Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu UNESP (HC-FMB/UNESP), Botucatu, São Paulo
  - Pontificia Universidade Catolica de Campinas (PUC-CAMP) - Hospital e Maternidade Celso Pierro (HMCP) - Centro de Pesquisa São Lucas, Campinas, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Conjunto Hospitalar de Mandaqui, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, São Paulo
  - Instituto Nacional de Infectologia Evandro Chagas / Fundação Oswaldo Cruz (FIOCRUZ), Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 3 countries (US, Brazil and Argentina). Participants were hospitalized with a confirmed lab PCR SARS-COV-2 infection.
  First Subject First Visit was on 26 May 2021 and Last Subject Last Visit was on 19May2022.
Pre-assignment Details: There were 223 participants screened for the study. Of these, 194 participants were randomized to received either asapiprant or placebo.
Groups:
- Asapiprant (BGE-175): Participants received two 50 mg tablets of asapiprant once daily for 14 days
- Placebo: Participants received two 50 mg tablets of matching placebo tablet daily for 14 days
Period: Overall Study
Arm/Group | Asapiprant (BGE-175) | Placebo
Started | 96 | 98
Completed | 78 | 87
Not Completed | 18 | 11
Not completed — Death | 16 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set includes all randomized participants and was used for baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Asapiprant (BGE-175) | Placebo | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Customized [Count of Participants; unit: Participants]
  Age 50 to less than 75 | 71 | 71 | 142
  Age greater or equal to 75 | 25 | 27 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 52 | 55 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 68 | 137
  Not Hispanic or Latino | 24 | 30 | 54
  Unknown or Not Reported | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Black or African American | 10 | 7 | 17
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 78 | 85 | 163
  Race: Other | 8 | 6 | 14
  Race: Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 21 | 21 | 42
  South America | 75 | 77 | 152
Baseline WHO ordinal scale [Count of Participants; unit: Participants] — WHO scale is as follows: 0) Uninfected 1) Ambulatory with no limitation of activities 2) Ambulatory with limitation of activities 3) Hospitalized, mild disease with no oxygen therapy 4) Hospitalized, mild disease with oxygen by mask or nasal prongs 5) Hospitalized, severe disease with noninvasive ventilation or high-flow oxygen 6) Hospitalized, severe disease with intubation and mechanical ventilation 7) Hospitalized, severe disease with ventilation and additional organ support (pressors, renal retention therapy, extracorporeal membrane oxygenation) 8) Death. Higher score means worse outcome.
  Participants
    WHO ordinal scale score 3 | 12 | 7 | 19
    WHO ordinal scale score 4 | 82 | 91 | 173
    WHO ordinal scale score 5 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Have Died or Progressed to Respiratory Failure
Description: Proportion of participants who have died or progressed to respiratory failure as defined by progressing to the need for high-flow nasal cannula O2 delivery, noninvasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) at Day 28.
  The proportion of participants is represented as a percentage.
Time Frame: First dose date up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set was used for the primary efficacy analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 94 | 97
Participants | 31 | 26
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.3312, Regression, Logistic; Odds Ratio (OR) = 1.366, 95% CI 2-sided [0.728 to 2.562]

2. Secondary Outcome: Proportion of Participants Experiencing Treatment-emergent Adverse Events
Description: Proportion of participants experiencing treatment-emergent adverse events as measured by the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
  The proportion of participants is represented as a percentage.
Time Frame: First dose of treatment through study Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 73 | 71

3. Secondary Outcome: Survival
Description: Proportion of participants surviving at Day 14, Day 28, and Day 57. The proportion of participants is represented as a percentage.
Time Frame: Baseline through Day 57; at Day 14, Day 28 and Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants. Subjects who discontinued the study prior to the timepoint are censored at the date of discontinuation and excluded from the analysis. At Day 57, the number participants analyzed were different because 9 participants were censored from the asapiprant arm and 15 participants from the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 94 | 96
Participants
  Survival at Day 14 | 89 | 93
  Survival at Day 28 | 79 | 87
  Survival at Day 57: number analyzed (Participants) | 85 | 81
  Survival at Day 57 | 69 | 72
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Day 14; Test type: Superiority; p = 0.4561, Regression, Logistic; Odds Ratio (OR) = 0.574, 95% CI 2-sided [0.133 to 2.475]
Statistical Analysis 2: Comparison: Asapiprant (BGE-175) vs Placebo; Day 28; Test type: Superiority; p = 0.1559, Regression, Logistic; Odds Ratio (OR) = 0.521, 95% CI 2-sided [0.212 to 1.282]
Statistical Analysis 3: Comparison: Asapiprant (BGE-175) vs Placebo; Day 57; Test type: Superiority; p = 0.1293, Regression, Logistic; Odds Ratio (OR) = 0.498, 95% CI 2-sided [0.203 to 1.226]

4. Secondary Outcome: Proportion of Subjects Who Survive Without Progression to Respiratory Failure Through Day 28
Description: Proportion of subjects who survive without progression to respiratory failure at Day 28.
  The proportion of participants is represented as a percentage.
Time Frame: First dose of treatment through Day 14, Day 28
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
percentage of participants
  Day 14 | 69.5 [59.1 to 77.7] | 78.6 [69.0 to 85.5]
  Day 28 | 67.3 [56.9 to 75.8] | 73.4 [63.4 to 81.0]
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Statistical analysis was only performed for Day 28. This is timeframe used for the primary endpoint; Test type: Superiority; p = 0.2687, Log Rank

5. Secondary Outcome: Time to Two Successive Negative Viral Titers in Nasopharyngeal Swabs
Description: Kaplan-Meier Estimate of Time to Two Successive Negative Viral Titers in Nasopharyngeal Swab (median)
Time Frame: Baseline through Day 28
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
days | 29 [29 to NA] — At Day 28, there were not enough events therefore the upper limit of 95% CI was unable to be calculated. | 29 [29 to NA] — At Day 28, there were not enough events therefore the upper limit of 95% CI was unable to be calculated.
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.3977, Log Rank

6. Secondary Outcome: Time to Clinical Worsening From Baseline Value (Defined by Time to ≥ 1-point Worsening on WHO Ordinal Scale for COVID-19)
Description: Kaplan-Meier Estimate of Time to Clinical Worsening from Baseline Value. Time to clinical worsening from baseline value (defined by time to ≥ 1-point worsening on World Health Organization (WHO) Ordinal Scale for COVID-19). The ordinal scale is an assessment of the clinical status at a given day. Each day, the worst score from the previous day will be recorded. The scale is as follows: 0.) Uninfected 1.) Ambulatory with no limitation of activities 2.) Ambulatory with limitation of activities 3.) Hospitalized, mild disease with no oxygen therapy 4.) Hospitalized, mild disease with oxygen by mask or nasal prongs 5.) Hospitalized, severe disease with noninvasive ventilation or high-flow oxygen 6.) Hospitalized, severe disease with intubation and mechanical ventilation 7.) Hospitalized, severe disease with ventilation and additional organ support (pressors, renal retention therapy, extracorporeal membrane oxygenation) 8.) Death. A higher score means a worse outcome.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
days | NA [NA to NA] — Median Survival Time was assessed using a Kaplan Meier Estimate with median survival defined as the smallest time at which the survival probability drops to 0.5 (50%) or below. Up to Day 57, the survival rate, for each of the treatment arms and overall, never fell below 50% therefore the median survival time was unable to be calculated. There were insufficient number of participants with events to calculate the lower limit of the 95% confidence interval. | NA [NA to NA] — Median Survival Time was assessed using a Kaplan Meier Estimate with median survival defined as the smallest time at which the survival probability drops to 0.5 (50%) or below. Up to Day 57, the survival rate, for each of the treatment arms and overall, never fell below 50% therefore the median survival time was unable to be calculated. There were insufficient number of participants with events to calculate the lower limit of the 95% confidence interval.
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.2229, Log Rank

7. Secondary Outcome: Proportion of Patients Who Develop Critical COVID-19 Illness
Description: Proportion of patients who develop critical COVID-19 illness as defined by at least one of the following:
  A. RF defined based on resource utilization requiring at least one of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, ECMO, clinical diagnosis respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation) B. Hemodynamic compromise (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressors) C. Multi-organ dysfunction/failure
  The proportion of participants is represented as a percentage.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 34 | 28
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.2941, Regression, Logistic; Odds Ratio (OR) = 1.388, 95% CI 2-sided [0.752 to 2.561]

8. Secondary Outcome: Time to Clinical Improvement From Baseline Value (Defined by Time to ≥ 1-point Improvement on WHO Ordinal Scale for COVID-19 Score - Must be Maintained Through Day 28)
Description: Kaplan-Meier Estimate of Time to Clinical Improvement from Baseline Value. Time to clinical improvement defined by time to ≥ 1-point improvement on World Health Organization (WHO) Ordinal Scale for COVID-19 - must be maintained through Day 28. The ordinal scale is an assessment of the clinical status at a given day. Each day, the worst score from the previous day will be recorded. The scale is as follows: 0.) Uninfected 1.) Ambulatory with no limitation of activities 2.) Ambulatory with limitation of activities 3.) Hospitalized, mild disease with no oxygen therapy 4.) Hospitalized, mild disease with oxygen by mask or nasal prongs 5.) Hospitalized, severe disease with noninvasive ventilation or high-flow oxygen 6.) Hospitalized, severe disease with intubation and mechanical ventilation 7.) Hospitalized, severe disease with ventilation and additional organ support (pressors, renal retention therapy, extracorporeal membrane oxygenation) 8.) Death. A higher score means a worse outcome.
Time Frame: First dose date up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
days | 8 [6.0 to 10.0] | 6 [5.0 to 9.0]
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.3325, Log Rank

9. Secondary Outcome: Mean Change From Baseline in WHO Ordinal Scale for COVID-19 Score
Description: Mean change from baseline in WHO Ordinal Scale for COVID-19 score
  World Health Organization (WHO) Ordinal Scale for COVID-19. The ordinal scale is an assessment of the clinical status at a given day. Each day, the worst score from the previous day will be recorded. The scale is as follows: 0.) Uninfected 1.) Ambulatory with no limitation of activities 2.) Ambulatory with limitation of activities 3.) Hospitalized, mild disease with no oxygen therapy 4.) Hospitalized, mild disease with oxygen by mask or nasal prongs 5.) Hospitalized, severe disease with noninvasive ventilation or high-flow oxygen 6.) Hospitalized, severe disease with intubation and mechanical ventilation 7.) Hospitalized, severe disease with ventilation and additional organ support (pressors, renal retention therapy, extracorporeal membrane oxygenation) 8.) Death. A higher score means a worse outcome.
Time Frame: Day 14/End of Treatment, Day 28, Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
score on a scale
  Change at Day 14 | -1.2 (2.17) | -1.8 (1.76)
  Change at Day 28 | -1.2 (2.51) | -1.7 (2.11)
  Change at Day 57: number analyzed (Participants) | 69 | 78
  Change at Day 57 | -2.7 (0.58) | -2.8 (0.42)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.0254, ANCOVA — Change at Day 14; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [0.08 to 1.2]
Statistical Analysis 2: Comparison: Asapiprant (BGE-175) vs Placebo; Change at Day 28; Test type: Superiority; p = 0.1109, ANCOVA; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.12 to 1.18]
Statistical Analysis 3: Comparison: Asapiprant (BGE-175) vs Placebo; Change at Day 57; Test type: Superiority; p = 0.8640, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.10 to 0.12]

10. Secondary Outcome: Number of Patients Who Had Intubation During the Study
Description: Proportion of Patients who had Intubation during the study defined as proportion of patients who had any documented intubation during the study.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 18 | 10
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.0919, Regression, Logistic; Odds Ratio (OR) = 2.046, 95% CI 2-sided [0.89 to 4.706]

11. Secondary Outcome: Duration of Intubation
Description: Duration of Intubation (first post-dosing intubation)
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 18 | 10
Days | 11.8 (5.32) | 7.8 (7.96)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.749, ANCOVA; Mean Difference (Final Values) = 3.83, 95% CI 2-sided [-0.42 to 8.08]

12. Secondary Outcome: Time to Discharge From Hospital Intensive Care Unit
Description: Time from intensive care unit admission to the recorded time of intensive care unit discharge
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 22 | 17
days | 15.7 (7.67) | 12.1 (8.55)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.1769, ANCOVA; Mean Difference (Final Values) = 3.69, 95% CI 2-sided [-1.75 to 9.13]

13. Secondary Outcome: Number of Patients Who Had Supplemental Oxygen Administration
Description: Proportion of patients who had any documented post-dosing supplemental O2 administration during the study.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 86 | 92
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.2621, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.184 to 1.586]

14. Secondary Outcome: Duration of Supplemental Oxygen Administration
Description: Duration of participants receiving supplemental oxygen
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 86 | 92
days | 14.7 (17) | 11.7 (14.81)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.2265, ANCOVA; Mean Difference (Final Values) = 2.81, 95% CI 2-sided [-1.76 to 7.37]

15. Secondary Outcome: Number of Patients Who Had Noninvasive Ventilation or High-flow Nasal Cannula O2 Administration
Description: Proportion of patients who had any documented post-dosing noninvasive ventilation or high-flow nasal cannula O2 administration.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 26 | 23
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.5497, Regression, Logistic; Odds Ratio (OR) = 1.223, 95% CI 2-sided [0.633 to 2.364]

16. Secondary Outcome: Duration of Noninvasive Ventilation by Nonrebreather Mask or High-flow Nasal Cannula
Description: Duration of participants receiving noninvasive ventilation by nonrebreather mask or high-flow nasal cannula
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 26 | 23
days | 11.1 (13.27) | 5.4 (7)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.1172, ANCOVA; Mean Difference (Final Values) = 4.89, 95% CI 2-sided [-1.27 to 11.05]

17. Secondary Outcome: Number of Patients Who Had Mechanical Ventilation.
Description: Proportion of patients who had any documented post-dosing mechanical ventilation.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
  This outcome is based on subjects who had WHO ordinal scale score of 6. A subject can have either a score of 6 or 7 (see outcome measure: Duration of Mechanical Ventilation Plus Additional Organ Support) but not both. This is the reason for the differing numbers for outcome 17 and 19.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 9 | 10
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.853, Regression, Logistic; Odds Ratio (OR) = 0.914, 95% CI 2-sided [0.353 to 2.368]

18. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of participants receiving mechanical ventilation
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 9 | 10
days | 10.9 (4.99) | 7.7 (4.88)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.1991, ANCOVA; Mean Difference (Final Values) = 3.16, 95% CI 2-sided [-1.86 to 8.18]

19. Secondary Outcome: Number of Patients Who Had Mechanical Ventilation Plus Additional Organ Support Using Vasopressors, and/or Renal Replacement Therapy and/or ECMO.
Description: Proportion of patients who had any documented post-dosing mechanical ventilation plus additional organ support using vasopressors, and/or renal replacement therapy and/or ECMO.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
  This outcome is based on subjects who had WHO ordinal scale score of 7. A subject can have either a score of 6 (see outcome measure: Duration of Mechanical Ventilation) or 7 but not both. This is the reason for the differing numbers for outcome 17 and 19.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 14 | 4
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.0166, Regression, Logistic; Odds Ratio (OR) = 4.103, 95% CI 2-sided [1.293 to 13.027]

20. Secondary Outcome: Duration of Mechanical Ventilation Plus Additional Organ Support Using Vasopressors, and/or Renal Replacement Therapy and/or ECMO
Description: Duration of participants receiving mechanical ventilation plus additional organ support using vasopressors, and/or renal replacement therapy and/or ECMO
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 14 | 4
days | 8.7 (5.85) | 3 (1.41)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.1297, ANCOVA; Mean Difference (Final Values) = 4.56, 95% CI 2-sided [-1.51 to 10.64]

21. Secondary Outcome: Daily Ratio of Oxygen Saturation (SpO2) to Fractional Inspired O2 (SpO2/FiO2)
Description: Daily ratio of participants' oxygen saturation (SpO2) to fractional inspired O2 (SpO2/FiO2)
Time Frame: First dose date up to Day 28
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: Ratio SpO2/FiO2
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Ratio SpO2/FiO2
  Baseline: number analyzed (Participants) | 65 | 75
  Baseline | 2.9 (0.71) | 3.0 (0.63)
  Treatment Day 2: number analyzed (Participants) | 69 | 76
  Treatment Day 2 | 2.7 (0.81) | 2.9 (0.73)
  Treatment Day 3: number analyzed (Participants) | 57 | 66
  Treatment Day 3 | 2.5 (0.92) | 2.8 (0.75)
  Treatment Day 4: number analyzed (Participants) | 48 | 50
  Treatment Day 4 | 2.3 (0.92) | 2.7 (0.86)
  Treatment Day 5: number analyzed (Participants) | 44 | 41
  Treatment Day 5 | 2.3 (0.91) | 2.6 (0.90)
  Treatment Day 6: number analyzed (Participants) | 40 | 35
  Treatment Day 6 | 2.3 (0.89) | 2.5 (0.90)
  Treatment Day 7: number analyzed (Participants) | 41 | 34
  Treatment Day 7 | 2.5 (0.99) | 2.6 (0.93)
  Treatment Day 8: number analyzed (Participants) | 36 | 31
  Treatment Day 8 | 2.4 (0.88) | 2.7 (0.95)
  Treatment Day 9: number analyzed (Participants) | 32 | 27
  Treatment Day 9 | 2.3 (1.02) | 2.8 (0.95)
  Treatment Day 10: number analyzed (Participants) | 31 | 24
  Treatment Day 10 | 2.3 (1.11) | 2.9 (0.67)
  Treatment Day 11: number analyzed (Participants) | 28 | 20
  Treatment Day 11 | 2.4 (1.10) | 2.8 (0.64)
  Treatment Day 12: number analyzed (Participants) | 24 | 19
  Treatment Day 12 | 2.2 (0.93) | 2.9 (0.72)
  Treatment Day 13: number analyzed (Participants) | 23 | 18
  Treatment Day 13 | 2.2 (0.71) | 2.8 (0.71)
  Treatment Day 14: number analyzed (Participants) | 24 | 18
  Treatment Day 14 | 2.2 (0.77) | 3.0 (0.73)
  Time of Discharge Visit: number analyzed (Participants) | 14 | 13
  Time of Discharge Visit | 3.1 (0.36) | 3.2 (0.42)
  Follow up Day 28: number analyzed (Participants) | 12 | 7
  Follow up Day 28 | 3.2 (0.44) | 3.0 (0.85)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Baseline; Test type: Superiority; p = 0.1916, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.35 to 0.07]
Statistical Analysis 2: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 2; Test type: Superiority; p = 0.1097, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.44 to 0.05]
Statistical Analysis 3: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 3; Test type: Superiority; p = 0.0276, ANCOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.63 to -0.04]
Statistical Analysis 4: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 4; Test type: Superiority; p = 0.0463, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.71 to -0.01]
Statistical Analysis 5: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 5; Test type: Superiority; p = 0.0969, ANCOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.71 to 0.06]
Statistical Analysis 6: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 6; Test type: Superiority; p = 0.4367, ANCOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.57 to 0.25]
Statistical Analysis 7: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 7; Test type: Superiority; p = 0.6685, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.54 to 0.35]
Statistical Analysis 8: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 8; Test type: Superiority; p = 0.2287, ANCOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.73 to 0.18]
Statistical Analysis 9: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 9; Test type: Superiority; p = 0.1061, ANCOVA; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.96 to 0.09]
Statistical Analysis 10: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 10; Test type: Superiority; p = 0.0415, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.06 to -0.02]
Statistical Analysis 11: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 11; Test type: Superiority; p = 0.1236, ANCOVA; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.00 to 0.12]
Statistical Analysis 12: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 12; Test type: Superiority; p = 0.0097, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.23 to -0.18]
Statistical Analysis 13: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 13; Test type: Superiority; p = 0.0157, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.02 to -0.11]
Statistical Analysis 14: Comparison: Asapiprant (BGE-175) vs Placebo; Treatment Day 14; Test type: Superiority; p = 0.0010, ANCOVA; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.32 to -0.36]
Statistical Analysis 15: Comparison: Asapiprant (BGE-175) vs Placebo; Time of Discharge Visit; Test type: Superiority; p = 0.6440, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.40 to 0.25]
Statistical Analysis 16: Comparison: Asapiprant (BGE-175) vs Placebo; Follow up Day 28; Test type: Superiority; p = 0.9869, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.60 to 0.59]

22. Secondary Outcome: Time to Discharge From the Hospital
Description: Length (in days) of the time of hospitalization until medical discharge
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
days | 10.8 (10.73) | 9.1 (9.09)
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.2399, ANCOVA; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-1.14 to 4.52]

23. Secondary Outcome: Number of Patients With Re-hospitalization
Description: Proportion of patients who are hospitalized again after the discharge of first hospitalization.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 6 | 7
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.8081, Regression, Logistic; Odds Ratio (OR) = 0.869, 95% CI 2-sided [0.28 to 2.695]

24. Secondary Outcome: Proportion of Participants Requiring Intensive Care Unit Admission
Description: Proportion of participants admitted to hospital intensive care unit post randomization.
  The proportion of participants is represented as a percentage.
Time Frame: First dose date up to Day 57
Population: The Intent-to-Treat (ITT) Analysis Set was used for the analysis and includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asapiprant (BGE-175) | Placebo
Number analyzed (Participants) | 96 | 98
Participants | 22 | 17
Statistical Analysis 1: Comparison: Asapiprant (BGE-175) vs Placebo; Test type: Superiority; p = 0.3193, Regression, Logistic; Odds Ratio (OR) = 1.436, 95% CI 2-sided [0.704 to 2.929]

ADVERSE EVENTS:
Time Frame: From first dose of treatment through Study Day 57
Groups:
- Asapiprant: Participants received two 50 mg tablets of asapiprant once daily for 14 days
Arm/Group | Asapiprant | Placebo
All-Cause Mortality (participants affected / at risk) | 16/96 | 10/98
Serious Adverse Events (participants affected / at risk) | 34/96 | 32/98
Other Adverse Events (participants affected / at risk) | 34/96 | 32/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asapiprant (N=96) | Placebo (N=98)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 21 (22)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 9 (9) | 4 (4)
Pulmonary sepsis (Infections and infestations) | 3 (4) | 4 (5)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 1 (3)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cardiac output decreased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asapiprant (N=96) | Placebo (N=98)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (8) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (8)
Constipation (Gastrointestinal disorders) | 15 (15) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 5 (6) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04705597/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04705597/SAP_001.pdf